CLINICAL TRIAL: NCT01247220
Title: REVOLUTIONARY: REtinal Vein OccLUsion Treatment With Scatter Laser Guided by Ultra Widefield angIOgraphy in combiNAtion With Ranibizumab Study Phase II
Brief Title: REtinal Vein OccLUsion Treatment With Scatter Laser Guided by UWFA in combiNAtion With Ranibizumab Study
Acronym: Revolution
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Retina Associates of Florida, P.A. (Other)
Responsible Party: Principal Investigator, Ivan J. Suner, MD, Director of Clinical Research, Retina Associates of Florida, P.A.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20101717
Record Dates: First submitted 2010-11-17; First posted 2010-11-24 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Macular Edema; Branch Retinal Vein Occlusion
Keywords: Macular Edema; Branch retinal vein occlusion; Ranibizumab
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Ranibizumab; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peripheral Laser + Ranibizumab (Experimental): Angiography-directed peripheral laser + ranibizumab
  Interventions: Drug: Ranibizumab; Procedure: Peripheral Laser
- Ranibizumab (Active Comparator): Ranibizumab
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal Ranibizumab 0.5 mg
  Other Names: Standard of Care; Intravitreal Anti-VEGF
Procedure: Peripheral Laser — Angiography-directed peripheral laser
  Other Names: Experimental; Scatter Laser
  Arms: Peripheral Laser + Ranibizumab

SUMMARY:
Branch retinal vein occlusion is a leading cause of vision loss. Treatment with ranibizumab (vascular endothelial growth factor (VEGF) inhibitor) on a monthly basis has been associated with improved vision results. There is a subgroup of patients with peripheral nonperfusion on ultrawidefield angiography that appears to be more dependent on anti-VEGF treatment.

In this trial the investigators compare the gold standard of monthly ranibizumab injections with ranibizumab + peripheral scatter laser to the areas of nonperfusion on angiography. Each group will have monthly injections for the first six months, then as needed by either visual acuity decrease or increased retinal thickness for the subsequent six months.

The primary outcome is visual acuity. Secondary outcomes are reduction in optical coherence tomography, and number of ranibizumab injections

DETAILED DESCRIPTION:
SUBJECTS Subject Selection Twenty subjects from a single site in the United States will be enrolled. Eligible subjects will have provided informed consent. (See Appendix A, the study flow chart, for screening assessments.)

Inclusion Criteria

Subjects will be eligible if the following criteria are met:

Ability to provide written informed consent and comply with study assessments for the full duration of the study Age > 18 years

Disease related considerations:

Study eye with macular edema secondary to branch retinal vein occlusion characterized by:

Fovea-involved macular edema of less than 12 months peripheral nonperfusion defined as at least 5 disc areas of contiguous nonperfusion on ultra-widefield fluorescein angiography absence of macular traction on clinical exam, UWFA, and OCT.

Study eye with best corrected visual acuity between 20/40 (≤ 73 letters on ETDRS chart) and 20/320 (≥ 19 letters on ETDRS chart) Other considerations Patient able to complete all study visits

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

Pregnancy (positive pregnancy test) or lactation. Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.

Prior enrollment in the study Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated Participation in another simultaneous medical investigation or trial Therapy with intravitreal triamcinolone, pegaptanib, ranibizumab, or bevacizumab within the previous 3 months Previous macular or panretinal scatter laser photocoagulation Previous pars plana vitrectomy Visually-significant significant cataracts as primary reason for vision loss Myocardial infarction or cerebrovascular accident within 6 months

METHOD OF TREATMENT ASSIGNMENT Patients meeting the study criteria and providing informed consent will be randomized according to the attached randomization chart (Appendix E) to study or control arm until 10 eyes are assigned to each group. Patients with both eyes eligible for the study will be assigned by coin flip.

STUDY TREATMENT Formulation Ranibizumab is formulated as a sterile solution aseptically filled in a sterile, 2 mL or 3-mL stoppered glass vial. Each single use vial is designed to deliver 0.05 mL of 10 mg/mL ranibizumab aqueous solution with 10 mM histidine HCI, 10%, trehalose dihydrate, and 0.01% polysorbate 20, pH 5.5. Each vial contains no preservative and is suitable for single use only.

Further details and molecule characterization will be included in the Investigator Brochure.

Dosage, Administration, and Storage

1. Dosage Patients in the treatment and control arms will receive intravitreal injection of 0.5 mg ranibizumab on the screening/Day 0 visit, and months 1 - 5. The need for subsequent injections at months 6 - 11 will be determined by presence of persistent or recurrent intraretinal fluid on OCT evaluation.
2. Administration
3. Storage Upon receipt, study drug kits should be refrigerated at 2C - 8C (36F - 46F). DO NOT FREEZE. Do not use beyond the expiration date. Ranibizumab vials should remain refrigerated. Protect vials from direct sunlight. Store in original carton until time of use.

   RANIBIZUMAB VIALS ARE FOR SINGLE USE ONLY. Vials used for one subject may not be used for any other subject.

   CONCOMITANT AND EXCLUDED THERAPIES Subjects may continue to receive all medications and standard treatments administered for their conditions at the discretion of their treating physician.

   STUDY ASSESSMENTS Assessments during the Treatment Period Screening / Day 0 Visit Informed consent Demographic data Medical and ocular history Vital signs (BP, heart rate) Pregnancy test (if applicable) Best corrected visual acuity (BCVA) ETDRS chart Slit lamp examination Intraocular pressure Dilated fundus examination Optical Coherence Tomography UWFA Ranibizumab treatment + peripheral laser tx (Treatment group) Ranibizumab treatment (Comparative group) SAE Monitoring Post-injection Phone Follow-up Update medical and ocular history SAE Monitoring Months 1, 2, 3, 4, and 5 Visits Update medical and ocular history Vital signs Best corrected visual acuity (BCVA) ETDRS chart Slit lamp examination Intraocular pressure Dilated fundus examination UWFA (Month 3) Ranibizumab treatment (Treatment and Comparative group) Optical Coherence Tomography SAE monitoring Month 6 Visit Update medical and ocular history Vital signs Best corrected visual acuity (BCVA) ETDRS chart Slit lamp examination Intraocular pressure Dilated fundus examination Optical Coherence Tomography UWFA SAE monitoring Months 6, 7, 8, 9, 10, 11, and 12 Visits Update medical and ocular history Vital signs Best corrected visual acuity (BCVA) ETDRS chart Slit lamp examination Intraocular pressure Dilated fundus examination Optical Coherence Tomography Ranibizumab treatment if necessary as determined by Optical Coherence Tomography assessment (Treatment and Comparative group) SAE monitoring

   Early Termination Assessments Subjects who withdraw from the study prior to completion should return for an early termination evaluation 30 days (14 days) following the last injection/study visit for monitoring of all adverse events (serious and nonserious). The schedule of assessments for early termination is the same as that for the final visit.

   SUBJECT DISCONTINUATION Subjects have a right to withdraw from the study at any time. The subject may be withdrawn from the study for any reasons: if it is in the best interest of the subject, intercurrent illness, adverse events, or worsening condition. The Western IRB may request the withdrawal of a subject because of protocol violations, administrative reasons, or any other valid and ethical reasons.

   If a subject discontinues from the study, he or she will not be allowed to re enter the study.

   Reasons for subject discontinuation may include, but are not limited to, the following:

   Sensory rhegmatogenous retinal detachment or Stage 3 or 4 macular hole Investigator determination that it is not in the best interest of the subject to continue participation Pregnancy Verteporfin PDT treatment in the study eye Pegaptanib sodium injection treatment in either eye Bevacizumab injection in either eye SAE Any other safety concerns In the event of an adverse event in the study eye that is considered by the investigator to be severe in intensity, serious consideration should be given to discontinuing the subject from the study.

   STUDY DISCONTINUATION

   This study may be terminated by Western IRB or Retina Associates of Florida at any time. Reasons for terminating the study may include the following:

   The incidence or severity of adverse events in this or other studies indicates a potential health hazard to subjects Subject enrollment is unsatisfactory Data recording is inaccurate or incomplete

   STATISTICAL METHODS Analysis of the Conduct of the Study There is no formal sample size calculation in this pilot study. As this is a phase I study, a sample size of 30 patients is chosen, making sure that it is feasible financially to conduct the study and logistically to complete the study within 18 months. If and when the study is planned for a phase II randomized control trial, appropriate statistical analysis will be determined.

   Safety Analyses Any adverse events, laboratory assessments, physical examinations, vital signs, ocular examinations and measurements from all 30 subjects will be utilized to summarize safety data for this pilot study.

   Efficacy Analyses Primary Endpoint Mean change in best corrected visual acuity (BCVA), as assessed by the number of letters read correctly on the ETDRS eye chart at a starting test distance of 4 meters at Month 6. This will also include eyes with gain of 15 letters or more, or loss of 15 letters or more on the ETDRS eye chart Secondary Endpoints Mean change in best corrected visual acuity (BCVA), as assessed by the number of letters read correctly on the ETDRS eye chart at a starting test distance of 4 meters at Month 2.

   Percent reduction of foveal thickness by optical coherence tomography. Percent reduction of macular volume by optical coherence tomography. Mean number of injections between Months 6 and 12.

   Missing Data Analyses of efficacy and safety will be based on available cases, without imputation for missing values.

   Interim Analyses No formal schedule of interim analyses is planned. Reports of adverse events from this study may be reviewed and summarized periodically while the study is ongoing to ensure the safety of subjects.

   DATA QUALITY ASSURANCE Accurate, consistent, and reliable data will be ensured through the use of standard practices and procedures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible if the following criteria are met:
* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years

  * Disease related considerations:
  * Study eye with macular edema secondary to branch retinal vein occlusion characterized by:
* Fovea-involved macular edema of less than 12 months peripheral nonperfusion defined as at least 5 disc areas of contiguous nonperfusion on ultra-widefield fluorescein angiography absence of macular traction on clinical exam, UWFA, and OCT.
* Study eye with best corrected visual acuity between 20/40 (≤ 73 letters on ETDRS chart) and 20/320 (≥ 19 letters on ETDRS chart)
* Other considerations
* Patient able to complete all study visits

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from this study:

  * Pregnancy (positive pregnancy test) or lactation. Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
  * Prior enrollment in the study
  * Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
  * Participation in another simultaneous medical investigation or trial
  * Therapy with intravitreal triamcinolone, pegaptanib, ranibizumab, or bevacizumab within the previous 3 months
  * Previous macular or panretinal scatter laser photocoagulation
  * Previous pars plana vitrectomy
  * Visually-significant significant cataracts as primary reason for vision loss
  * Myocardial infarction or cerebrovascular accident within 6 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan J Suner, MD, Study Chair — Retina Associates of Florida, P.A.
Locations (1):
- Retina Associates of Florida, P.A., Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peripheral Laser + Ranibizumab | Ranibizumab
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peripheral Laser + Ranibizumab | Ranibizumab | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (18) | 70 (10) | 69.5 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: ETDRS visual acuity
Time Frame: 6 and 12 months
Measure: Mean (Standard Deviation); unit: letters on ETDRS Visual Acuity Chart
Arm/Group | Peripheral Laser + Ranibizumab | Ranibizumab
Number analyzed (Participants) | 6 | 6
letters on ETDRS Visual Acuity Chart
  6 month results | 16.8 (10.1) | 14.5 (11.6)
  12 month results | 19.1 (7.4) | 15.3 (13.2)

2. Secondary Outcome: Number of Ranibizumab Injections
Description: Number of ranibizumab injections needed by decreased visual acuity and/or increasing retinal thickness in second six months of observation period
Time Frame: 12 months
Measure: Mean (Full Range); unit: injections
Arm/Group | Peripheral Laser + Ranibizumab | Ranibizumab
Number analyzed (Participants) | 6 | 6
injections | 0.06 [0 to 1] | 2.2 [1 to 4]

3. Secondary Outcome: Retinal Thickness
Description: central foveal thickness on optical coherence tomography
Time Frame: 6 and 12 months
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Peripheral Laser + Ranibizumab | Ranibizumab
Number analyzed (Participants) | 6 | 6
microns
  6 month results | 207 (47) | 241 (45)
  12 month results | 282 (26) | 281 (29)

ADVERSE EVENTS:
Arm/Group | Peripheral Laser + Ranibizumab | Ranibizumab
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
small study size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No